CLINICAL TRIAL: NCT05228717
Title: Point-of-care Lung Ultrasound (POCUS)-Integrated Observation Study of Admitted Patients With COVID-19
Brief Title: Point-of-care Lung Ultrasound (POCUS)-Integrated Study of Admitted Patients With COVID-19
Acronym: PIOS-COVID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Olive View-UCLA Education & Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 1590419
Record Dates: First submitted 2021-03-10; First posted 2022-02-08 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Lung Injury; ARDS; Acute Cardiac Event; Covid19; Ultrasound; Hypoxemia; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Lung Injury; COVID-19; Hypoxia; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID+: Patients with confirmed COVID-19 pneumonia as the primary diagnosis, or COVID-associated acute hypoxemic respiratory failure or hypoxia (minimum O2 requirement 3L), that are being admitted from the emergency department, who either have waiver of consent, give verbal consent to participate, or have NOK (next of kin) provide consent.
  Exclusion criteria: age <18 years old, pregnant patients, or patients that verbally refuse participation Intervention/observation: q48-72h POCUS of the lungs, heart, and IVC
  Interventions: Diagnostic Test: Point of Care Ultrasound

INTERVENTIONS:
Diagnostic Test: Point of Care Ultrasound — q48-72h point of care ultrasound of the lungs, heart, and IVC (inferior vena cava)

SUMMARY:
This study seeks to define the ultrasound profile of patients with COVID-19, and document the progression of these ultrasound findings to develop prognostication and clinical decision instruments that can help guide management of patient with COVID-19. Primary aims include the development of ARDS, refractory hypoxemia, acute cardiac injury, pulmonary embolism, pneumothorax or death. Secondary aims include potential change in CT and plain film utilization given the use of POCUS, as well as emergency department and inpatient LOS (length of stay).

DETAILED DESCRIPTION:
A. SPECIFIC AIMS

1. To define the lung ultrasound profile of patients admitted with COVID-19 pneumonia, hypoxia, or hypoxemic respiratory failure.
2. To document the progression of POCUS findings in admitted patients with COVID-19 respiratory failure.
3. Along with other clinical data, to develop a prognostication and clinical decision instrument that can help guide management of patients with COVID-19, specifically for the following specific outcomes:

   * Development of ARDS, worsening oxygen requirement, or need for intubation. On POCUS, this would be associated with a shift in lateral lung involvement to anterior lung zone involvement; or overall increase in B-lines for all lung zones
   * Refractory hypoxemia requiring lung recruitment maneuvers, including prone positioning or ECMO (extra-corporeal membrane oxygenation). On POCUS, this would be associated with the presence of posterior-lateral alveolar consolidation, which gives the appearance of "hepatization of lung"
   * Development of acute cardiac injury, as defined by acute coronary syndrome or myocarditis. On POCUS, this would be associated with the development of worsening systolic function
   * Development of pulmonary embolism as defined by CT evidence, +DVT (deep vein thrombosis), or therapeutic anticoagulation. On POCUS, this would be associated with a RV (right ventricle) strain pattern (D-shaped septum on parasternal short axis, RV>LV (left ventricle) diameter on apical)
   * Development of pneumothorax. On POCUS, this would be associated with the absence of pleural sliding

   A composite outcome of development of ARDS, acute cardiac injury, hypoxemic respiratory failure requiring prone positioning or ECMO, PE (pulmonary embolism), PTX (pneumothorax), or death, will be used as the primary outcome.

   These are secondary aims that investigators will assess, but not base our power calculation on:
4. To assess the potential change of using POCUS in CT and plain film utilization, as well as emergency department and inpatient LOS.
5. If current triage workflow related to the COVID-19 pandemic integrates POCUS into triage, investigators will extend this analysis to the point of triage, and not just admitted patients.
6. To assess the prevalence of lung ultrasound findings suggestive of COVID-19 infection in patients that present with acute coronary syndromes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed COVID-19 pneumonia as the primary diagnosis, or COVID- associated acute hypoxemic respiratory failure or hypoxia (minimum O2 requirement 3L), that are being admitted from the emergency department, who either have waiver of consent, give verbal consent to participate, or have next of kin give consent for participation.

Exclusion Criteria:

* age < 18 years old, pregnant patients, or patients that verbally refuse participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients with COVID-19 Pneumonia/hypoxemic respiratory failure requiring at least 3L of O2.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2020-11-10 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Association of POCUS changes with major clinical events | From admission to 21 days, or endpoint reached
  Association of POCUS worsening with development of a composite outcome of development of ARDS, acute cardiac injury, hypoxemic respiratory failure requiring prone positioning or ECMO, pneumothorax, cardiac tamponade, or death.
Time from POCUS worsening to clinical diagnosis. | From admission to 21 days, or endpoint reached
  Time interval from POCUS worsening to clinical diagnosis. Investigators will measure the duration between POCUS worsening and clinical diagnosis of any of the major clinical events described in outcome 1.

SECONDARY OUTCOMES:
Utilization of traditional radiography | From admission to 21 days, or endpoint reached
  To assess the potential change of using POCUS in CT and plain film utilization, as well as emergency department and inpatient LOS.
Individual clinical outcomes | From admission to 21 days, or endpoint reached
  Investigators will compare POCUS changes and the time interval to development of each of the following outcomes: ARDS, acute cardiac injury, hypoxemic respiratory failure requiring prone positioning or ECMO, pneumothorax, cardiac tamponade, or death.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - UCLA-Ronald Reagan, Los Angeles, California
  - Olive View-UCLA, Sylmar, California
  - SUNY Downstate, New York, New York
  - Temple University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ai T, Yang Z, Hou H, Zhan C, Chen C, Lv W, Tao Q, Sun Z, Xia L. Correlation of Chest CT and RT-PCR Testing for Coronavirus Disease 2019 (COVID-19) in China: A Report of 1014 Cases. Radiology. 2020 Aug;296(2):E32-E40. doi: 10.1148/radiol.2020200642. Epub 2020 Feb 26. PMID 32101510
- [Background] Bouhemad B, Brisson H, Le-Guen M, Arbelot C, Lu Q, Rouby JJ. Bedside ultrasound assessment of positive end-expiratory pressure-induced lung recruitment. Am J Respir Crit Care Med. 2011 Feb 1;183(3):341-7. doi: 10.1164/rccm.201003-0369OC. Epub 2010 Sep 17. PMID 20851923
- [Background] Buonsenso D, Pata D, Chiaretti A. COVID-19 outbreak: less stethoscope, more ultrasound. Lancet Respir Med. 2020 May;8(5):e27. doi: 10.1016/S2213-2600(20)30120-X. Epub 2020 Mar 20. No abstract available. PMID 32203708
- [Background] Chavez MA, Shams N, Ellington LE, Naithani N, Gilman RH, Steinhoff MC, Santosham M, Black RE, Price C, Gross M, Checkley W. Lung ultrasound for the diagnosis of pneumonia in adults: a systematic review and meta-analysis. Respir Res. 2014 Apr 23;15(1):50. doi: 10.1186/1465-9921-15-50. PMID 24758612
- [Background] Cheng Z, Lu Y, Cao Q, Qin L, Pan Z, Yan F, Yang W. Clinical Features and Chest CT Manifestations of Coronavirus Disease 2019 (COVID-19) in a Single-Center Study in Shanghai, China. AJR Am J Roentgenol. 2020 Jul;215(1):121-126. doi: 10.2214/AJR.20.22959. Epub 2020 Mar 14. PMID 32174128
- [Background] Chung M, Bernheim A, Mei X, Zhang N, Huang M, Zeng X, Cui J, Xu W, Yang Y, Fayad ZA, Jacobi A, Li K, Li S, Shan H. CT Imaging Features of 2019 Novel Coronavirus (2019-nCoV). Radiology. 2020 Apr;295(1):202-207. doi: 10.1148/radiol.2020200230. Epub 2020 Feb 4. PMID 32017661
- [Background] Clerkin K, Fried J, Raikhelkar J, et al. Coronavirus Disease 2019 (COVID-19) and Cardiovascular Disease. Circulation. 2020 Mar 21. doi: 10.1161/CIRCULATIONAHA.120.046941.
- [Background] Copetti R, Soldati G, Copetti P. Chest sonography: a useful tool to differentiate acute cardiogenic pulmonary edema from acute respiratory distress syndrome. Cardiovasc Ultrasound. 2008 Apr 29;6:16. doi: 10.1186/1476-7120-6-16. PMID 18442425
- [Background] Dietrich CF, Mathis G, Cui XW, Ignee A, Hocke M, Hirche TO. Ultrasound of the pleurae and lungs. Ultrasound Med Biol. 2015 Feb;41(2):351-65. doi: 10.1016/j.ultrasmedbio.2014.10.002. PMID 25592455
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Hasan AA, Makhlouf HA. B-lines: Transthoracic chest ultrasound signs useful in assessment of interstitial lung diseases. Ann Thorac Med. 2014 Apr;9(2):99-103. doi: 10.4103/1817-1737.128856. PMID 24791173
- [Background] Henderson WR, Griesdale DE, Dominelli P, Ronco JJ. Does prone positioning improve oxygenation and reduce mortality in patients with acute respiratory distress syndrome? Can Respir J. 2014 Jul-Aug;21(4):213-5. doi: 10.1155/2014/472136. Epub 2014 Jun 13. PMID 24927376
- [Background] Lichtenstein D, Goldstein I, Mourgeon E, Cluzel P, Grenier P, Rouby JJ. Comparative diagnostic performances of auscultation, chest radiography, and lung ultrasonography in acute respiratory distress syndrome. Anesthesiology. 2004 Jan;100(1):9-15. doi: 10.1097/00000542-200401000-00006. PMID 14695718
- [Background] Lichtenstein DA, Lascols N, Meziere G, Gepner A. Ultrasound diagnosis of alveolar consolidation in the critically ill. Intensive Care Med. 2004 Feb;30(2):276-281. doi: 10.1007/s00134-003-2075-6. Epub 2004 Jan 13. PMID 14722643
- [Background] Mayo PH, Beaulieu Y, Doelken P, Feller-Kopman D, Harrod C, Kaplan A, Oropello J, Vieillard-Baron A, Axler O, Lichtenstein D, Maury E, Slama M, Vignon P. American College of Chest Physicians/La Societe de Reanimation de Langue Francaise statement on competence in critical care ultrasonography. Chest. 2009 Apr;135(4):1050-1060. doi: 10.1378/chest.08-2305. Epub 2009 Feb 2. PMID 19188546
- [Background] Mayo PH, Copetti R, Feller-Kopman D, Mathis G, Maury E, Mongodi S, Mojoli F, Volpicelli G, Zanobetti M. Thoracic ultrasonography: a narrative review. Intensive Care Med. 2019 Sep;45(9):1200-1211. doi: 10.1007/s00134-019-05725-8. Epub 2019 Aug 15. PMID 31418060
- [Background] Pan F, Ye T, Sun P, Gui S, Liang B, Li L, Zheng D, Wang J, Hesketh RL, Yang L, Zheng C. Time Course of Lung Changes at Chest CT during Recovery from Coronavirus Disease 2019 (COVID-19). Radiology. 2020 Jun;295(3):715-721. doi: 10.1148/radiol.2020200370. Epub 2020 Feb 13. PMID 32053470
- [Background] Peng QY, Wang XT, Zhang LN; Chinese Critical Care Ultrasound Study Group (CCUSG). Findings of lung ultrasonography of novel corona virus pneumonia during the 2019-2020 epidemic. Intensive Care Med. 2020 May;46(5):849-850. doi: 10.1007/s00134-020-05996-6. Epub 2020 Mar 12. No abstract available. PMID 32166346
- [Background] Silva S, Biendel C, Ruiz J, Olivier M, Bataille B, Geeraerts T, Mari A, Riu B, Fourcade O, Genestal M. Usefulness of cardiothoracic chest ultrasound in the management of acute respiratory failure in critical care practice. Chest. 2013 Sep;144(3):859-865. doi: 10.1378/chest.13-0167. PMID 23670087
- [Background] Soldati G, Smargiassi A, Inchingolo R, Buonsenso D, Perrone T, Briganti DF, Perlini S, Torri E, Mariani A, Mossolani EE, Tursi F, Mento F, Demi L. Is There a Role for Lung Ultrasound During the COVID-19 Pandemic? J Ultrasound Med. 2020 Jul;39(7):1459-1462. doi: 10.1002/jum.15284. Epub 2020 Apr 7. No abstract available. PMID 32198775
- [Background] Soni NJ, Franco R, Velez MI, Schnobrich D, Dancel R, Restrepo MI, Mayo PH. Ultrasound in the diagnosis and management of pleural effusions. J Hosp Med. 2015 Dec;10(12):811-6. doi: 10.1002/jhm.2434. Epub 2015 Jul 28. PMID 26218493
- [Background] Sperandeo M, Filabozzi P, Varriale A, Carnevale V, Piattelli ML, Sperandeo G, Brunetti E, Decuzzi M. Role of thoracic ultrasound in the assessment of pleural and pulmonary diseases. J Ultrasound. 2008 Jun;11(2):39-46. doi: 10.1016/j.jus.2008.02.001. Epub 2008 Mar 17. PMID 23396553
- [Background] Stefanidis K, Dimopoulos S, Kolofousi C, Cokkinos DD, Chatzimichail K, Eisen LA, Wachtel M, Karakitsos D, Nanas S. Sonographic lobe localization of alveolar-interstitial syndrome in the critically ill. Crit Care Res Pract. 2012;2012:179719. doi: 10.1155/2012/179719. Epub 2012 May 9. PMID 22645669
- [Background] Volpicelli G, Elbarbary M, Blaivas M, Lichtenstein DA, Mathis G, Kirkpatrick AW, Melniker L, Gargani L, Noble VE, Via G, Dean A, Tsung JW, Soldati G, Copetti R, Bouhemad B, Reissig A, Agricola E, Rouby JJ, Arbelot C, Liteplo A, Sargsyan A, Silva F, Hoppmann R, Breitkreutz R, Seibel A, Neri L, Storti E, Petrovic T; International Liaison Committee on Lung Ultrasound (ILC-LUS) for International Consensus Conference on Lung Ultrasound (ICC-LUS). International evidence-based recommendations for point-of-care lung ultrasound. Intensive Care Med. 2012 Apr;38(4):577-91. doi: 10.1007/s00134-012-2513-4. Epub 2012 Mar 6. PMID 22392031
- [Background] Wu C, Chen X, Cai Y, Xia J, Zhou X, Xu S, Huang H, Zhang L, Zhou X, Du C, Zhang Y, Song J, Wang S, Chao Y, Yang Z, Xu J, Zhou X, Chen D, Xiong W, Xu L, Zhou F, Jiang J, Bai C, Zheng J, Song Y. Risk Factors Associated With Acute Respiratory Distress Syndrome and Death in Patients With Coronavirus Disease 2019 Pneumonia in Wuhan, China. JAMA Intern Med. 2020 Jul 1;180(7):934-943. doi: 10.1001/jamainternmed.2020.0994. PMID 32167524
- [Background] Young BE, Ong SWX, Kalimuddin S, Low JG, Tan SY, Loh J, Ng OT, Marimuthu K, Ang LW, Mak TM, Lau SK, Anderson DE, Chan KS, Tan TY, Ng TY, Cui L, Said Z, Kurupatham L, Chen MI, Chan M, Vasoo S, Wang LF, Tan BH, Lin RTP, Lee VJM, Leo YS, Lye DC; Singapore 2019 Novel Coronavirus Outbreak Research Team. Epidemiologic Features and Clinical Course of Patients Infected With SARS-CoV-2 in Singapore. JAMA. 2020 Apr 21;323(15):1488-1494. doi: 10.1001/jama.2020.3204. PMID 32125362
- [Background] Zhao W, Zhong Z, Xie X, Yu Q, Liu J. Relation Between Chest CT Findings and Clinical Conditions of Coronavirus Disease (COVID-19) Pneumonia: A Multicenter Study. AJR Am J Roentgenol. 2020 May;214(5):1072-1077. doi: 10.2214/AJR.20.22976. Epub 2020 Mar 3. PMID 32125873
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076